CLINICAL TRIAL: NCT00476346
Title: Calcium and Vitamin D Supplementation Decreases Incidence of Stress Fractures in Female Navy Recruits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: GlaxoSmithKline (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Joan M. Lappe, Creighton University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DAMD-17-01-1-0807
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2008-08

CONDITIONS: Stress Fracture
Keywords: physical training; military training; bone; fracture prevention; young adult
MeSH Terms: conditions — Fractures, Stress | interventions — Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calcium (Active Comparator): Daily calcium supplementation Intervention: Calcium 2000mg / daily
  Interventions: Dietary Supplement: Calcium & Vitamin D
- Vitamin D (Experimental): Daily Calcium and Vitamin D supplementation Intervention: Vitamin D 800IU / daily
  Interventions: Dietary Supplement: Calcium & Vitamin D

INTERVENTIONS:
Dietary Supplement: Calcium & Vitamin D — Calcium 2000mg / daily Vitamin D 800IU / daily

SUMMARY:
We conducted a double-blind, placebo-controlled randomized clinical trial of calcium and vitamin D supplementation in 5201 female Naval recruits. During 8 weeks of basic training, supplementation with 2000 mg calcium and 800 IU vitamin D/day decreased incidence of stress fracture by 25%. The hypothesis was:

Supplementation with calcium 2000 mg/d and vitamin D 800 IU/d will significantly reduce the incidence of stress fractures in female Navy recruits during 8 weeks of basic training.

DETAILED DESCRIPTION:
Introduction: Stress fractures (SFx) are one of the most common and debilitating overuse injuries seen in military recruits, and they are also problematic for non-military athletic populations. The goal of this randomized double-blind, placebo-controlled study was to determine if a calcium and vitamin D intervention could reduce the incidence of SFx in female recruits during basic training.

Methods: We recruited 5201 female Navy recruit volunteers and randomized them to a 2000 mg calcium and 800 IU vitamin D supplement/day or placebo. SFx were ascertained when recruits reported to the Great Lakes clinic with symptoms. All SFx were confirmed with radiography or technetium scan according to the usual Navy protocol.

Results: A total of 309 subjects were diagnosed with a SFx resulting in an incidence of 5.9% per eight weeks. Using "intention-to-treat" analysis by including all enrolled subjects, Fisher's Exact test found that the calcium and vitamin D group had a 25% lower incidence of SFx than the control group (6.6% vs 5.3%, respectively, p=0.03). The per protocol analysis, including only the 3700 recruits who completed the study, found a 27% lower incidence of fractures in the supplemented vs the control group (8.6% vs 6.8%, respectively, p=0.02).

Conclusions: Generalizing the findings to the population of 14,416 females who entered basic training at the Great Lakes during the 24 months of recruitment, calcium and vitamin D supplementation for the entire cohort would have prevented about 130 persons per year from fracturing. Such a decrease in SFx would be associated with a significant decrease in morbidity and financial costs.

ELIGIBILITY:
Inclusion Criteria:

* Female entering basic recruit training at the Great Lakes Naval Station

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5201 (Actual)
Dates: Start 2002-05; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
individuals with stress fracture | one year

CONTACTS AND LOCATIONS:
Overall Officials: Joan M Lappe, Ph.D., Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States